CLINICAL TRIAL: NCT04210284
Title: Oral Nutritional Optimization in Total Joint Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-01976
Record Dates: First submitted 2019-12-23; First posted 2019-12-24 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutritional supplementation (Experimental): Given Ensure Max Protein Nutrition shake 2 weeks before surgery and continued 2 weeks after surgery.
  Interventions: Dietary Supplement: Ensure
- No Nutritional supplementation (No Intervention): Treatment as usual

INTERVENTIONS:
Dietary Supplement: Ensure — Ensure Max Protein Shake is an over the counter available drinkable nutritional supplement. Per serving, it contains:
  * 160 Calories, 20 from fat
  * 2g Total fat
  * 0.5g Saturated fat
  * 20mg Cholesterol
  * 135mg Sodium
  * 170mg Potassium
  * 19g Total carbohydrate
  * <1g Fiber
  * 4g Sugar
  * 16g Protein
  Participants will receive Ensure High Protein for 2 weeks pre- and 4 weeks post-operatively. These patients will be instructed to consume 1 serving (16fl oz) of Ensure High Protein daily. They will be provided with this product at a pre-operative clinical visit or have it mailed to their home. Hematologic nutritional values will be measured as specified previously.
  Descriptive statistics will be used to report baseline characteristics and primary study objectives. Hematologic outcomes will be compared between the control ("NO ENSURE") and oral supplementation ("ENSURE") arms for the aforementioned baseline and perioperative variables
  Arms: Nutritional supplementation

SUMMARY:
The purpose of this study is to determine the effect on hematological markers of nutritional intervention on nutritionally deficient patients following total joint replacement surgery.

DETAILED DESCRIPTION:
Numerous pre-operative modifiable variables have been extensively investigated for their effect on outcomes in TJA. These include metabolic diseases such as diabetes mellitus, obesity, and smoking status. However, nutritional status has not been as thoroughly investigated; to date, no prospective randomized control study has assessed the effect of oral nutritional supplementation for malnourished patients. This study will be a novel investigation into the role for routine serum screening for malnutrition as well as oral nutritional supplementation in TJA patients. This study could serve as a stepping stone towards creating a new pathway to highlight at-risk patients and pre-operatively optimizing their outcomes after TJA.

ELIGIBILITY:
Inclusion Criteria:

1. Patient are current candidates for elective primary total hip and total knee arthroplasty
2. Patients ≥55 years of age but ≤ 95
3. Patients who meet at least one of the following three laboratory criteria for malnutrition:

TSerum Albumin: ≤3.5 mg/dl Pre-Albumin: <15 mg/dl Transferrin: <200 mg/dl

Exclusion Criteria:

1. Previous history of septic arthritis
2. Allergy to oral supplementation
3. Inability to consume oral supplementation
4. Protein malabsorption syndromes
5. Eating disorders
6. End stage renal and hepatic disease
7. Revision surgery, non-elective surgery, hemiarthroplasty, and unicompartmental knee arthroplasty

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-07-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in the patients' albumin, pre-albumin, and/or transferrin levels | Visit 2 (2 wks pre) Visit 3 (surgery day) Visit 5 (4 weeks post)
  Biological specimen collection and laboratory evaluations- all included patients' hematologic markers of malnutrition (albumin, pre-albumin, and transferrin) will be recorded at 2 weeks prior to surgery, the day of surgery, and 6 weeks. These blood tests can all be performed from one sample of blood at each visit. The results will then be accessed via the EMR

CONTACTS AND LOCATIONS:
Overall Officials: Ran Schwarzkopf, Principal Investigator — NYU Langone
Locations (2):
- United States (2):
  - NYU Langone Health, New York, New York
  - Rothman Orthopedic Institute, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data. Upon reasonable request Requests should be directed to Daniel.waren@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.